CLINICAL TRIAL: NCT05033106
Title: Comparison Between Intravitreal Injection of Ranibizumab and Bevacizumab for Treatment of Type 1 Retinopathy of Prematurity
Brief Title: Ranibizumab Vs Bevacizumab for Type 1 Retinopathy of Prematurity
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zagazig University (Other Government)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Ghada Mahmoud Tawfik Ibrahim Eladawy, dr_ghadaeladawy@yahoo.com, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D-9-2020
Record Dates: First submitted 2021-08-26; First posted 2021-09-02 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Retinopathy of Prematurity Both Eyes
MeSH Terms: interventions — Bevacizumab; Ranibizumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eyes with IVI bevacizumab (Active Comparator): 0.625 mg/0.025 mL bevacizumab is injected into the vitreous cavity of the left eye
  Interventions: Drug: Bevacizumab, Ranibizumab
- Eyes with IVI ranibizumab (Active Comparator): A dose of 0.25 mg/0.025 mL ranibizumab (Lucentis) is injected in the right eye of the infant
  Interventions: Drug: Bevacizumab, Ranibizumab

INTERVENTIONS:
Drug: Bevacizumab, Ranibizumab — • A dose of 0.25 mg/0.025 mL ranibizumab (Lucentis) is injected in the right eye of the infant and 0.625 mg/0.025 mL bevacizumab is injected into the vitreous cavity of the left eye 1 mm posterior to the superior/inferior temporal limbus via 30 G needle. The two injections are done sequentially on two consecutive days starting with the eye of more advanced disease.
  Other Names: avastin, leucentis

SUMMARY:
Retinopathy of prematurity (ROP) with inadequate growth and development of retinal blood vessels in premature infants is one of the foremost reasons for childhood blindness. Recently there is a shift of treatment to VEGF inhibitors which can regress ROP without destroying the peripheral retina. Yet, the best drug has not been identified.Bevacizumab is a larger, full-length immunoglobulin G (IgG) molecule with slower retinal clearance and therefore prolonged diffusion into the systemic circulation, up to 3 weeks. In contrast, the systemic half-life of a Fab molecule, such as ranibizumab, is a few hours. The objective is to compare the efficacy and reliability of intravitreal bevacizumab with standard 0.625 mg dose and intravitreal ranibizumab treatments for type 1 ROP, namely pattern of disease regression, recurrence of ROP, necessity of subsequent ablative procedures.

DETAILED DESCRIPTION:
Objectives

To compare the efficacy and reliability of intravitreal bevacizumab with standard 0.625 mg dose and intravitreal ranibizumab treatments for type 1 ROP, namely pattern of disease regression, recurrence of ROP, necessity of subsequent ablative procedures.

Study population & Sample size Infants with Type 1 ROP (affecting both eyes) screened at neonatal intensive care unit (NICU) of Cairo University.

The sample size is calculated to be 36 eyes of 18 infants using open Epi confidence total 95%, power of the study 80% according to the following : the mean SD of axial length of patients with stage 3 ROP using bevacizumab versus ranibizumab (20.3 1.16 versus 19.4 ).

Study Design

This is a prospective, comparative, interventional non inferiority study.

Methods

* Infants with type 1 ROP affecting both eyes will be included.
* Before intravitreal injection, the parents or legal guardian of the infants will be informed about the procedure.
* After written consent is obtained, the pupil will be dilated with 2.5% phenylephrine and 0.5% tropicamide injection.
* The injections will be performed in the operating theatre under general (light inhalational anesthesia) or topical anesthesia with Benoxinate hydrochloride 0.4%.
* Povidone iodine10% swab will be applied on the eyelids and eyelashes. A sterile eyelid speculum will be inserted. Each eye will be meticulously bathed with 5% povidone iodine solution for 3 min before intravitreal injection.
* A dose of 0.25 mg/0.025 mL ranibizumab (Lucentis) is injected in the right eye of the infant and 0.625 mg/0.025 mL bevacizumab is injected into the vitreous cavity of the left eye 1 mm posterior to the superior/inferior temporal limbus via 30 G needle. The two injections are done sequentially on two consecutive days starting with the eye of more advanced disease.
* Fundus examination will be conducted with an indirect ophthalmoscope and a 28-D lens. The central retinal artery and the lens will be evaluated in addition to whether a retinal tear is present.
* Postoperative moxifloxacin 0.4% drops will be prescribed 4 times daily for one week.
* Patients will be seen 24 hours after first injection, to monitor for any signs of infection.
* Infants will then be seen weekly for 4 weeks and dilated fundus examination and and digital coloured fundus images by RetCam will be performed to document response of the disease.
* Success criteria to the IVB injection will be defined as, during the follow up period of 60 weeks' postmenstrual age:

  * recovery of the plus disease
  * regression of any stage of ROP
  * progression of peripheral retinal vascularization
* If any progression occurs in the disease course, in terms of: increase in plus disease or progression to higher stage of ROP, immediate second IVB dose 0.625mg will be given to either groups.
* Follow-up will be continued for a minimum of one year corrected age or until we ensure complete peripheral retinal vascularization.

ELIGIBILITY:
Inclusion Criteria:

- Infants with a birth weight of ≤ 1500 g or geststional age of ≤ 30 weeks and selected infants with birth weight between 1500 and 2000 g or gestational age of more than 30 weeks with an unstable clinical course, including those requiring cardiorespiratory support. Patients with bilateral disease who will receive bilateral injections, are only included. Type 1 ROP according to ETROP study which is defined as, Zone I ROP with plus disease, Zone I, stage 3 ROP without plus disease and Zone II, stage 2 or 3 ROP with plus disease.

Exclusion Criteria:

Eyes with previous intravitreal injections. Eyes with previous laser therapy. Eyes with any other pathology, other than ROP. Eyes with ROP stage 4 or 5. Eyes with mucopurulent or purulent conjunctivitis. Infants who will not be able to comply to the follow-up schedule.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
• Regression achieved either by single injection or multiple injections or additional laser therapy at 60 weeks postmenstrual age. | 60 weeks PMA
  regression of plus disease and the active neovessels

SECONDARY OUTCOMES:
• Recurrence of ROP | 60 weeks PMA
  (recurrent plus disease, recurrent neovascularization, or reformation of ridge despite treatment)

OTHER OUTCOMES:
• The number and kind of adverse events, the number of patients progressing to stage 4 or 5. | 60 weeks PMA
  stage 4, retinal detachment and stage 5,cicatricial ROP
• The number of reinjections or laser spots and the number of eyes that need lensectomy and vitrectomy. | 60 weeks PMA
  reinjection with anti-VEGF, or indirect laser
• Refractive errors in spherical equivalent in patients who only received anti-VEGF treatment, pattern of fixation and ocular alignment. | 60 weeks PMA
  Retinoscopy is done to detect errors of refraction

CONTACTS AND LOCATIONS:
Overall Officials: Ghada Mahmoud Tawfik Eladawy, Msc, Principal Investigator — Zagazig University
Locations (1):
- Zagazig University, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: Yes
International Publishing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: two years
Access Criteria: Internet